CLINICAL TRIAL: NCT03400709
Title: Protective Role of N-acetylcisteine From Cisplatin-induced Ototoxicity in Patients With Head and Neck Cancer. A Randomized, Placebo Controlled Clinical Trial
Brief Title: Protective Role of N-acetylcisteine From Cisplatin-induced Ototoxicity in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Juan de Dios, Santiago (Other)
Responsible Party: Principal Investigator, Daniel Munoz MD, MSc., Otolaryngologist, Clinical Epidemiologist., Hospital San Juan de Dios, Santiago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 123606
Record Dates: First submitted 2017-12-27; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Cisplatin Adverse Reaction; Hearing Loss Ototoxic
Keywords: Cisplatin; Ototoxicity; N-acetylcisteine
MeSH Terms: conditions — Ototoxicity | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetylcisteine group (Experimental)
  Interventions: Drug: N Acetylcysteine
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: N Acetylcysteine — Oral administration of drug, before, during and after Chemoradiotherapy including Cisplatin.
  Arms: N-acetylcisteine group
Drug: Placebo Oral Tablet — Placebo treatment
  Arms: Control group

SUMMARY:
Introduction. Cisplatin-induced ototoxicity is a very frequent event and its consequences can cause a lot of deterioration in patients. Early diagnosis is essential because it would allow the appropriate implementation of strategies to reduce its effect. Among these N-acetylcysteine, an antioxidant agent that has shown otoprotective effect. Study design. Randomized, parallel design and placebo controlled clinical trial. Methods. Patients with head and neck cancer who require treatment with cisplatin were enrolled in 2 branches: a control group that receives a placebo and experimental group that receives the drug. High-frequency audiometries (6 - 16 KHz) are performed before, during and after the treatment finalization.

ELIGIBILITY:
Inclusion Criteria:

* Adults Patients with Head and Neck Squamous Cell carcinoma requiring Chemoradiotherapy including Cisplatin.

Exclusion Criteria:

* Conductive Hearing Loss
* SNHL with >= 40db PTA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Hearing threshold | Baseline.
  High frequencies pure tone average
Hearing threshold | up to 4th week of chemoradiotherapy
  High frequencies pure tone average
Hearing threshold | through study completion, an average of 3 months
  High frequencies pure tone average

CONTACTS AND LOCATIONS:
Locations (1):
- Daniel Munoz, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No